CLINICAL TRIAL: NCT07203547
Title: Multicenter, Randomized, Double-blind, Active Control, Parallel, Non-inferior, Phase 4 Clinical Trial to Assess Efficacy and Safety of Laybon Tab. in Patients With Knee Osteoarthritis
Brief Title: Phase 4 Study of Laybon Tab. in Knee Osteoarthritis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mather's Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MTS-RAY-401
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis
Keywords: Laybon Tab.; Knee Osteoarthritis; Osteoarthritis; OA; Non-inferiority; Randomized Trial; Double blind; Phase 4
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants, investigators, and study staff are blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Drug Group (Experimental)
  Interventions: Drug: Laybon Tab.
- Control Drug Group (Active Comparator)
  Interventions: Drug: Layla Tab.

INTERVENTIONS:
Drug: Layla Tab. — Layla Tab., oral, twice daily, 8 weeks.
  Arms: Control Drug Group
Drug: Laybon Tab. — Laybon Tab., oral, twice daily, 8 weeks.
  Arms: Test Drug Group

SUMMARY:
This Phase 4, multicenter, randomized, double-blind, active-controlled, parallel study aims to evaluate the non-inferiority of Laybon Tab. compared to Layla Tab. (PMG Pharm Co., Ltd.) in patients with knee osteoarthritis. Participants will receive either Laybon Tab. or Layla Tab. for 8 weeks. The primary outcome is the change in knee pain during activity, assessed by a 100 mm pain VAS over the previous 24 hours.

DETAILED DESCRIPTION:
This phase 4 clinical trial will assess the efficacy and safety of Laybon Tab. compared to Layla Tab. in adults with knee osteoarthritis. Participants will be randomized in a double-blind, parallel, active-controlled design to receive either Laybon Tab. or Layla Tab. for 8 weeks. The primary endpoint is the change in activity-related knee pain over the past 24 hours, measured by a 100 mm visual analogue scale (VAS). Secondary endpoints include additional efficacy and safety evaluations. The study aims to demonstrate the non-inferiority of Laybon Tab. to Layla Tab. All participants will be monitored for efficacy, safety, and medication compliance, and standard eligibility criteria will be applied.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 40 to 80 years, male or female.
2. Diagnosed with unilateral or bilateral knee osteoarthritis according to the American College of Rheumatology (ACR) clinical criteria, meeting at least 3 of the following:

   * Age > 50 years
   * Morning stiffness < 30 minutes
   * Crepitus
   * Bony tenderness
   * Bony enlargement
   * No warmth on palpation
3. Knee osteoarthritis pain persisting for at least 3 months and requiring pharmacologic treatment at screening.
4. Kellgren-Lawrence grade 1-3 on knee X-ray at screening.
5. Knee pain during activity over the past 24 hours ≤ 80 mm on 100 mm pain VAS at screening.
6. Knee pain during activity over the past 24 hours ≥ 40 mm on 100 mm pain VAS at baseline (Visit 2).
7. Able to walk without assistance (walker, cane, etc.). Participants who have routinely used mobility aids for at least 6 months prior to screening may continue their usual aid throughout the study.
8. Women of childbearing potential and men must agree to use medically acceptable contraception during the study, including hormonal contraception, IUD/IUS, bilateral tubal ligation, partner vasectomy, or sexual abstinence.
9. Participants currently receiving treatment for knee osteoarthritis must agree to discontinue prior therapies and comply with a wash-out period before and during study participation
10. Participants must have received and understood a full explanation of the study and voluntarily provided written informed consent.
11. Women of childbearing potential must have a negative pregnancy test prior to study drug administration.

Exclusion Criteria:

1. Screening BMI ≥ 35.0 kg/m².
2. Presence of other joint disorders or systemic conditions that could affect safety or efficacy assessments, including:

   * Rheumatoid arthritis, autoimmune diseases, septic arthritis, inflammatory joint diseases, gout, recurrent pseudogout, joint fracture, ochronosis, acromegaly, hemochromatosis, Wilson's disease, primary osteochondrodysplasia, genetic disorders (e.g., hypermobility), or secondary osteoarthritis
   * Severe osteoarthritis of hip or other joints interfering with knee evaluation
   * Painful conditions such as Sudeck's atrophy, Paget's disease, spinal disc herniation
   * Active or suspected infection in the target knee
3. History of the following conditions at screening:

   * Upper gastrointestinal ulcer within 6 months, GI bleeding within 12 months, or gastrointestinal disorders affecting drug absorption
   * Severe cardiovascular diseases (NYHA class ≥3, ischemic heart disease, arrhythmia, peripheral vascular disease, prior coronary interventions, cerebrovascular disorders)
   * Severe liver impairment (ALT or AST > 3× ULN)
   * Severe renal impairment (eGFR < 30 mL/min)
   * Bronchial asthma
   * Fluid retention
   * Lipid metabolism disorders (hyperlipidemia, diabetic dyslipidemia, pancreatitis)
   * Active systemic infection or viral infection (HCV, HBV)
   * Malignancy, except those in complete remission ≥5 years or certain completely treated cancers (basal cell carcinoma, squamous cell carcinoma, thyroid papillary carcinoma, cervical carcinoma in situ)
4. Current use of psychotropic medications.
5. History of knee interventions prior to study drug administration:

   * Cell or gene therapy, autologous bone marrow stem cell therapy within 5 years
   * Knee ligament surgery, cartilage graft, osteotomy within 1 year
   * Arthroscopy within 6 months
   * Intra-articular injections (HA, PN, PDRN, PRP, collagen, dextrose/prolotherapy) within 6 months
   * Steroid injections, other anti-inflammatory injections, unknown knee medications within 3 months
   * Continuous opioid use ≥1 week within 3 months
   * Systemic steroids (excluding inhaled) or anticonvulsants within 1 month
   * Prior knee joint replacement
6. Individuals who have received the following medications or therapies for the purpose of controlling pain or improving symptoms in the knee joint or other conditions prior to study drug administration and who are unable to discontinue these treatments during participation in the clinical trial, or who have additional treatments planned. (However, subjects may participate in the study after a 2-week wash-out period prior to study drug administration [Visit 2]. Low-dose aspirin up to 100 mg per day is permitted; the use of acetaminophen provided as rescue medication is allowed within the permitted dose, except within 48 hours prior to Visits 3 and 4.)

   * Acetaminophen, non-steroidal anti-inflammatory drugs (NSAIDs), and other analgesics.
   * Topical anti-inflammatory drugs for knee application (NSAID gel, cream, patch, etc.) or topical analgesics (including muscle pain relievers containing capsaicin, menthol, camphor, etc.).
   * Other therapies (e.g., physical therapy, oriental medicine such as acupuncture, cupping, and moxibustion).
   * Nutritional supplements for osteoarthritis (e.g., glucosamine, chondroitin, methylsulfonylmethane [MSM], boswellia, etc.).
7. Known hypersensitivity to study drug or rescue medications or their components.
8. History of allergy or hypersensitivity to COX-2 inhibitors, sulfonamides, aspirin, or other NSAIDs.
9. Pregnant or breastfeeding women.
10. Known allergy or hypersensitivity to soybean oil.
11. Known allergy or hypersensitivity to peanuts or legumes.
12. History of drug or alcohol abuse within 1 year prior to study drug administration.
13. High-risk alcohol consumption (≥2 times/week and ≥7 drinks per occasion for men, ≥5 for women).
14. Prior use of Layla Tab., Laybon Tab., or any herbal/extract product containing the same components (e.g., 25% ethanol extract of listed herbs) within the past 4 weeks (wash-out required).
15. Participation in another clinical trial or use of investigational medical device within 1 month prior to screening.
16. Unable to understand or provide informed consent as judged by the investigator.
17. Any other reason the investigator considers the participant unsuitable for study participation.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Knee Pain During Activity (100 mm Pain VAS) | Baseline and Week 8
  Change from baseline (Visit 2, prior to study drug administration) to Week 8 in activity-related knee pain over the past 24 hours, as assessed by a 100 mm pain Visual Analogue Scale (VAS).

SECONDARY OUTCOMES:
Change From Baseline in Knee Pain During Activity (100 mm Pain VAS) at Week 4 | Baseline and Week 4
  Change from baseline (Visit 2) to Week 4 in activity-related knee pain over the past 24 hours, assessed by 100 mm pain VAS.
Change From Baseline in WOMAC Total Score | Baseline, week 4 and week 8
  Change from baseline (Visit 2) to Week 4 and Week 8 in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) total score.
Change From Baseline in WOMAC Subscale Scores | Baseline, Week 4, and Week 8
  Change from baseline (Visit 2) to Week 4 and Week 8 in WOMAC subscale scores: pain, stiffness, and physical function.
Patient Global Assessment of Knee Osteoarthritis | Week 4 and Week 8
  Patient's global assessment of overall knee osteoarthritis symptoms using a 5-Point Likert Scale at Week 4 and Week 8.
Quality of Life Assessment Using SF-36 | Week 4 and Week 8
  Change in health-related quality of life measured by the SF-36 questionnaire at Week 4 and Week 8.
Use of Rescue Medication | Week 4 and Week 8
  Frequency and total amount of rescue medication used during the 8-week treatment period, evaluated at Week 4 and Week 8.

IPD SHARING:
Plan to Share IPD: No